CLINICAL TRIAL: NCT01662791
Title: Weight Loss in Parkinson's Disease and the Potential Role of Small Bowel Bacterial Overgrowth
Brief Title: Weight Loss in Parkinson's Disease and Role of Small Bowel Bacterial Overgrowth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John K. DiBaise, MD, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-006817
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Small Bowel Bacterial Overgrowth; Weight Loss; Gastrointestinal; Rifaximin
MeSH Terms: conditions — Parkinson Disease; Weight Loss | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case Group (Experimental): All individuals in the Case group (i.e., only the subjects who had lost weight) were offered open-label treatment with the poorly absorbed antibiotic, rifaximin, 550 mg PO twice a day (BID) for 14 days. Subjects in the case group were in the study for 3 months.
  Interventions: Drug: Rifaximin
- Control Group (No Intervention): This arm consisted of subjects with Parkinson's Disease who had not experienced significant weight loss. These patients were in the study for one day.

INTERVENTIONS:
Drug: Rifaximin — All individuals in the weight loss group (i.e., only the Case group) were offered open-label treatment with the poorly absorbed antibiotic, rifaximin, 550 mg PO BID for 14 days. Treatment will not depend upon the results of the bacterial overgrowth breath test. Thus, both normal and abnormal breath test subjects received antibiotic treatment.
  Other Names: Xifaxan
  Arms: Case Group

SUMMARY:
The potential role of small bowel bacterial overgrowth (SBBO) in weight loss occurring in patients with Parkinson's Disease (PD) has not previously been examined. Our hypothesis was that SBBO is an important contributor to the development of weight loss in individuals with PD. The investigators proposed to 1) examine the role of SBBO in weight loss occurring in patients with PD and 2) determine the response to its treatment with a poorly absorbed antibiotic. The investigators performed a prospective, observational case-control study (Part 1) with an open-label therapeutic component (Part 2). Cases were defined as those PD patients who experienced significant weight loss while Controls were defined as those PD patients who did not experience significant weight loss.

DETAILED DESCRIPTION:
Part 1:

Consecutive patients seen in the Parkinson's disease clinic at Mayo Clinic in Arizona were approached to participate. After the determination of their eligibility and appropriate signed informed consent, all PD patients (i.e., both Case and Control groups) underwent the following:

1. Assessment of demographic features, weight history and PD history
2. PD and other medications
3. Determination of PD severity using the Unified Parkinson's Disease rating scale
4. Gastrointestinal Symptom Severity Index (GISSI) and modified GISSI.
5. Determination of usual calorie and nutrient intake (Brief Block Food Frequency Questionnaire)
6. Paffenbarger physical activity questionnaire
7. Quality of life (SF12 and PD-specific)
8. Hospital Anxiety and Depression Scale
9. Glucose hydrogen breath test (SBBO test)
10. Qualitative assessments of smell and taste

All questionnaires were completed during the 2 hour breath test.

Part 2:

All individuals in the weight loss group (i.e., only the Case group) were offered open-label treatment with the poorly absorbed antibiotic, rifaximin, 550 mg PO twice a day for 14 days. Treatment did not depend upon the results of the bacterial overgrowth breath test. Thus, both normal and abnormal breath test subjects could have received antibiotic treatment. The patient was contacted by phone 1 month after treatment at which time the presence of GI symptoms was determined and inquiry made about any adverse effects related to rifaximin use. GI symptoms, quality of life, weight measurement, and breath testing were repeated at a 3 month study visit.

ELIGIBILITY:
Inclusion criteria: Parkinson's Disease

Exclusion Criteria:

1. Wheelchair-bound, akinetic individuals
2. Tube-fed individuals
3. Presence of dementia
4. Unwilling or unable to complete the tests
5. Allergic or intolerant to rifaximin
6. Presence of chronic upper or lower gastrointestinal disorders that have symptoms that may be confused with SBBO (e.g., irritable bowel syndrome, inflammatory bowel disease, celiac disease, functional dyspepsia, gastroparesis, and chronic pancreatitis)
7. Presence of prior surgery on the gastrointestinal tract except cholecystectomy, appendectomy or herniorrhaphy
8. Presence of severe concomitant acute or chronic medical condition that may interfere with the completion or interpretation of the test results
9. Women of childbearing potential. Given the age of patients with Parkinson's disease, we do not anticipate this being a large population.
10. Use of antibiotics within 1 month of breath testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Di Baise, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the Mayo Clinic in Scottsdale, Arizona.
Groups:
- Case Group: All individuals in the Case group (i.e., only the subjects who had lost weight) were offered open-label treatment with the poorly absorbed antibiotic, rifaximin, 550 mg PO twice a day (BID) for 14 days. Subjects in the case group were in the study for 3 months.
  Rifaximin: All individuals in the weight loss group (i.e., only the Case group) were offered open-label treatment with the poorly absorbed antibiotic, rifaximin, 550 mg PO BID for 14 days. Treatment did not depend upon the results of the bacterial overgrowth breath test. Thus, both normal and abnormal breath test subjects received antibiotic treatment.
- Control Group: This arm consisted of subjects with Parkinson's Disease who had not experienced significant weight loss. These patients were in the study for one day; they did not take part in the second part of the study.
Period: Part 1 - Observational
Arm/Group | Case Group | Control Group
Started | 8 | 41
Completed | 8 | 41
Not Completed | 0 | 0
Period: Part 2 - Interventional
Arm/Group | Case Group | Control Group
Started | 8 | 0 (The Control Group did not take part in the second part of the study.)
Completed | 8 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Case Group: All individuals in the Case group (i.e., only the subjects who had lost weight) were offered open-label treatment with the poorly absorbed antibiotic, rifaximin, 550 mg PO BID for 14 days. Subjects in the case group were in the study for 3 months.
  Rifaximin: All individuals in the weight loss group (i.e., only the Case group) were offered open-label treatment with the poorly absorbed antibiotic, rifaximin, 550 mg PO BID for 14 days. Treatment did not depend upon the results of the bacterial overgrowth breath test. Thus, both normal and abnormal breath test subjects received antibiotic treatment.
- Total: Total of all reporting groups
Arm/Group | Case Group | Control Group | Total
Number analyzed (Participants) | 8 | 41 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 11 | 11
  >=65 years | 8 | 30 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 17 | 19
  Male | 6 | 24 | 30
Region of Enrollment [Number; unit: participants]
  United States | 8 | 41 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Small Bowel Bacterial Overgrowth (SBBO)
Description: SBBO is measured by the Hydrogen Breath Test, which measures the hydrogen and methane gas produced by bacteria in the small bowel that has diffused into the blood, then lungs for expiration. After an overnight fast, subjects ingested a solution consisting of 50 grams of glucose mixed in 150 mL of water. Immediately before ingestion of glucose and at 20-minute intervals for 2 hours following ingestion, laboratory staff collected end-expiratory breath samples and analyzed them for hydrogen and methane using a Quintron sample correction (SC) breath microlyzer. A diagnosis of SBBO was defined by an increase in expiration of 12 parts per million (ppm) or more of hydrogen and/or methane.
Time Frame: Baseline to 2 hours
Measure: Number; unit: participants
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 8 | 41
participants
  12 ppm increase | 2 | 12
  20 ppm increase | 2 | 9
Statistical Analysis 1: Comparison: Case Group vs Control Group; Comparison between the groups for >12 ppm; Test type: Superiority or Other; p = 1.0, Chi-squared

2. Secondary Outcome: PD-specific Quality of Life Questionnaire (PDQ-39)
Description: The PDQ-39 is designed to address aspects of functioning and well-being for those affected by Parkinson's disease. This questionnaire is based on a multi-dimensional model of health. Eight subscale scores may be derived from the items: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognitions (4 items), communication (3 items), bodily discomfort (3 items). Patients are asked to think about their health and general well-being and to consider how often in the last month they have experienced certain events (e.g. difficulty walking 100 yards). Patients are asked to indicate the frequency of each event by selecting one of 5 options (Likert Scale): Never/occasionally/sometimes/often/always or cannot do at all. Each dimension is calculated as a scale from 0 to 100, with 0= no problem at all; 100= maximum level of problem. Sub-scale score are averaged to calculate the summary index.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 8 | 41
units on a scale
  Mobility | 23.1 (20.1) | 14.0 (17.6)
  Activities of Daily Living | 25.0 (14.1) | 18.1 (13.3)
  Emotional Well-Being | 17.2 (23.5) | 13.2 (11.5)
  Stigma | 13.3 (25.5) | 6.2 (9.9)
  Social Support | 3.1 (6.2) | 1.4 (4.9)
  Cognition | 32.0 (31.4) | 17.5 (12.8)
  Communication | 25.0 (27.1) | 10.8 (13.3)
  Bodily Discomfort | 24.0 (22.9) | 27.0 (22.7)
  Summary Index | 20.3 (19.3) | 13.5 (9.0)
Statistical Analysis 1: Comparison: Case Group vs Control Group; Comparison between groups for mobility sub-scale; Test type: Superiority or Other; p = 0.235, Chi-squared
Statistical Analysis 2: Comparison: Case Group vs Control Group; Comparison between groups for activities of daily living sub-scale; Test type: Superiority or Other; p = 0.206, Chi-squared
Statistical Analysis 3: Comparison: Case Group vs Control Group; Comparison between groups for emotional well-being sub-scale; Test type: Superiority or Other; p = 0.641, Chi-squared
Statistical Analysis 4: Comparison: Case Group vs Control Group; Comparison between groups for stigma sub-scale; Test type: Superiority or Other; p = 0.446, Chi-squared
Statistical Analysis 5: Comparison: Case Group vs Control Group; Comparison between groups for social support sub-scale; Test type: Superiority or Other; p = 0.466, Chi-squared
Statistical Analysis 6: Comparison: Case Group vs Control Group; Comparison between groups for cognition sub-scale; Test type: Superiority or Other; p = 0.205, Chi-squared
Statistical Analysis 7: Comparison: Case Group vs Control Group; Comparison between groups for communication sub-scale; Test type: Superiority or Other; p = 0.153, Chi-squared
Statistical Analysis 8: Comparison: Case Group vs Control Group; Comparison between groups for bodily discomfort sub-scale; Test type: Superiority or Other; p = 0.730, Chi-squared
Statistical Analysis 9: Comparison: Case Group vs Control Group; Comparison between groups for summary index sub-scale; Test type: Superiority or Other; p = 0.334, Chi-squared

3. Secondary Outcome: PD-specific Quality of Life Questionnaire (PDQ-39) Over Time in Case Group
Description: as for outcome 2
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 8 | 0
units on a scale
  Mobility baseline | 23.1 (20.1) |
  Mobility 3 months | 27.8 (25.5) |
  Activities of Daily Living baseline | 25.0 (14.1) |
  Activities of Daily Living 3 months | 17.7 (17.8) |
  Emotional Well-Being baseline | 17.2 (23.5) |
  Emotional Well-Being 3 months | 11.0 (22.9) |
  Stigma baseline | 13.3 (25.5) |
  Stigma 3 months | 5.5 (11.3) |
  Social Support baseline | 3.1 (6.2) |
  Social Support 3 months | 3.1 (6.2) |
  Cognition baseline | 32.0 (31.4) |
  Cognition 3 months | 21.9 (16.7) |
  Communication baseline | 25.0 (27.1) |
  Communication 3 months | 15.6 (10.4) |
  Bodily Discomfort baseline | 24.0 (22.9) |
  Bodily Discomfort 3 months | 30.2 (31.2) |
  Summary Index baseline | 20.3 (19.3) |
  Summary Index 3 months | 16.6 (13.3) |
Statistical Analysis 1: Comparison: Case Group; Comparison in case group between baseline and 3 months for mobility sub-scale; Test type: Superiority or Other; p = 0.167, McNemar
Statistical Analysis 2: Comparison: Case Group vs Control Group; Comparison in case group between baseline and 3 months for activities of daily living sub-scale; Test type: Superiority or Other; p = 0.159, McNemar
Statistical Analysis 3: Comparison: Case Group; Comparison in case group between baseline and 3 months for emotional well-being sub-scale; Test type: Superiority or Other; p = 0.041, McNemar
Statistical Analysis 4: Comparison: Case Group; Comparison in case group between baseline and 3 months for stigma sub-scale; Test type: Superiority or Other; p = 0.190, McNemar
Statistical Analysis 5: Comparison: Case Group; Comparison in case group between baseline and 3 months for social support sub-scale; Test type: Superiority or Other; p = 1.0, McNemar
Statistical Analysis 6: Comparison: Case Group; Comparison in case group between baseline and 3 months for cognition sub-scale; Test type: Superiority or Other; p = 0.160, McNemar
Statistical Analysis 7: Comparison: Case Group; Comparison in case group between baseline and 3 months for communication sub-scale; Test type: Superiority or Other; p = 0.276, McNemar
Statistical Analysis 8: Comparison: Case Group; Comparison in case group between baseline and 3 months for bodily discomfort sub-scale; Test type: Superiority or Other; p = 0.351, McNemar
Statistical Analysis 9: Comparison: Case Group; Comparison in case group between baseline and 3 months for summary index sub-scale; Test type: Superiority or Other; p = 0.186, McNemar

4. Secondary Outcome: Gastrointestinal Symptom Severity Index (GISSI)
Description: The GISSI is a validated, self-administered, multi-dimensional instrument designed to measure the frequency, severity and bothersomeness of individual GI symptoms and to provide subscale scores for interrelated symptom clusters. Factor analyses yielded 5 distinct symptom clusters that were labeled as Constipation/Difficult defecation; Abdominal Pain/Discomfort; Dyspepsia; Diarrhea/Fecal incontinence; Gastroesophageal reflux disease (GERD)/Chest symptoms; and Nausea/Vomiting. Scores could range from 0 to 100, with a higher score indicating greater severity of symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 8 | 41
units on a scale
  Constipation | 22.6 (20.8) | 14.5 (15.8)
  Dyspepsia | 7.2 (11.5) | 4.5 (6.6)
  Abdominal Pain/Discomfort | 8.1 (16.5) | 6.6 (10.2)
  Diarrhea | 3.4 (4.9) | 2.7 (6.2)
  GERD | 5.6 (10.6) | 3.4 (5.2)
  Nausea/Vomiting | 1.6 (3.1) | 0.63 (2.4)
Statistical Analysis 1: Comparison: Case Group vs Control Group; Comparison between groups for constipation sub-scale; Test type: Superiority or Other; p = 0.303, Chi-squared
Statistical Analysis 2: Comparison: Case Group vs Control Group; Comparison between groups for dyspepsia sub-scale; Test type: Superiority or Other; p = 0.518, Chi-squared
Statistical Analysis 3: Comparison: Case Group vs Control Group; Comparison between groups for abdominal discomfort sub-scale; Test type: Superiority or Other; p = 0.800, Chi-squared
Statistical Analysis 4: Comparison: Case Group vs Control Group; Comparison between groups for diarrhea sub-scale; Test type: Superiority or Other; p = 0.736, Chi-squared
Statistical Analysis 5: Comparison: Case Group vs Control Group; Comparison between groups for GERD sub-scale; Test type: Superiority or Other; p = 0.570, Chi-squared
Statistical Analysis 6: Comparison: Case Group vs Control Group; Comparison between groups for nausea and vomiting sub-scale; Test type: Superiority or Other; p = 0.394, Chi-squared

5. Secondary Outcome: Gastrointestinal Symptom Severity Index (GISSI) Over Time in Case Group
Description: as for outcome 4
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 8 | 0
units on a scale
  Constipation baseline | 32.3 (29.8) |
  Constipation 3 months | 10.0 (10.6) |
  Dyspepsia baseline | 12.9 (20.6) |
  Dyspepsia 3 months | 8.2 (15.5) |
  Abdominal Pain/Discomfort baseline | 14.5 (29.4) |
  Abdominal Pain/Discomfort 3 months | 4.0 (7.5) |
  Diarrhea baseline | 6.0 (8.7) |
  Diarrhea 3 months | 12.7 (19.8) |
  GERD baseline | 10.0 (18.9) |
  GERD 3 months | 8.5 (12.9) |
  Nausea/Vomiting baseline | 5.8 (11.1) |
  Nausea/Vomiting 3 months | 2.2 (6.3) |
Statistical Analysis 1: Comparison: Case Group; Comparison in case group between baseline and 3 months for constipation sub-scale; Test type: Superiority or Other; p = 0.056, McNemar
Statistical Analysis 2: Comparison: Case Group; Comparison in case group between baseline and 3 months for dyspepsia sub-scale; Test type: Superiority or Other; p = 0.380, McNemar
Statistical Analysis 3: Comparison: Case Group; Comparison in case group between baseline and 3 months for abdominal discomfort sub-scale; Test type: Superiority or Other; p = 0.244, McNemar
Statistical Analysis 4: Comparison: Case Group; Comparison in case group between baseline and 3 months for diarrhea sub-scale; Test type: Superiority or Other; p = 0.279, McNemar
Statistical Analysis 5: Comparison: Case Group; Comparison in case group between baseline and 3 months for GERD sub-scale; Test type: Superiority or Other; p = 0.554, McNemar
Statistical Analysis 6: Comparison: Case Group; Comparison in case group between baseline and 3 months for nausea and vomiting sub-scale; Test type: Superiority or Other; p = 0.351, McNemar

6. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: The HADS is a self-administered 14-item questionnaire (seven for anxiety and seven for depression) Items are rated on a 4-point scale from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. The cut-offs used for identifying significant psychiatric distress was >/= 8. This assessment was only measured at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 8 | 41
units on a scale
  Depression | 3.5 (3.7) | 3.3 (2.1)
  Anxiety | 3.8 (3.8) | 4.0 (2.6)
Statistical Analysis 1: Comparison: Case Group vs Control Group; Comparison between the two groups at baseline for depression; Test type: Superiority or Other; p = 0.872, t-test, 1 sided
Statistical Analysis 2: Comparison: Case Group vs Control Group; Comparison between the two groups at baseline for anxiety; Test type: Superiority or Other; p = 0.835, t-test, 1 sided

7. Other Pre Specified Outcome: Calories Consumed From Brief Block Food Frequency Questionnaire (FFQ)
Description: The FFQ is a validated, self-administered semi-quantitative questionnaire used to assess differences in macronutrient, and energy intake. It was designed to provide estimates of usual and customary dietary intake. This questionnaire contains a food list of about 70 food items.
  A Food Frequency Questionnaire (FFQ) is a limited checklist of foods and beverages with a frequency response section for subjects to report how often each item was consumed over a specified period of time. Semi-quantitative FFQs collect portion size information as standardized portions or as a choice of portion sizes. Calculations for nutrient intake or calories can be estimated via computerized software programs that multiply the reported frequency of each food by the amount of nutrient or calories in a serving of that food.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Calories
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 8 | 41
Calories
  Total calories consumed | 1503.7 (395.6) | 1588.0 (538.7)
  Fat | 36.3 (9.6) | 38.0 (6.5)
  Saturated Fat | 12.7 (3.8) | 13.0 (3.0)
  Protein | 13.4 (3.1) | 15.7 (3.4)
  Carbohydrate | 45.1 (7.6) | 43.7 (6.9)
  Alcohol | 14.8 (9.3) | 12.5 (8.8)
  Sweets | 10.9 (15.3) | 6.5 (7.1)

8. Secondary Outcome: Weight Change in Case Group After Treatment
Description: Weight change after treatment
Time Frame: baseline, 3 months
Measure: Number; unit: participants
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 8 | 0
participants
  Subjects who lost weight from baseline | 3 |
  Subjects who gained weight from baseline | 5 |

9. Secondary Outcome: Paffenbarger Physical Activity Questionnaire (PPAQ)
Description: The PPAQ is a validated, self-administered questionnaire that asks for a recall of physical activity of physical activity over the previous 1-week. From the answers to the questions, a physical activity index (PAI) can be computed, providing an estimate of energy expenditure in kcal/week.
  The PAI can be estimated using a list of the physical activities a person performs within a time period and the amount of time spent on each activity, e.g. walking to work, light housework, swimming, carrying bricks at work, or whatever applies to an individual person. There is a value called the physical activity ratio for each activity. The list of activities is used to find the relevant values of physical activity ratios, then an overall physical activity level value for the time period is calculated, using time-weighted averages of the physical activity ratios.
  This assessment was only measured at baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kcal/week
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 8 | 41
kcal/week | 848.8 (566.5) | 2253 (2027)

ADVERSE EVENTS:
Arm/Group | Case Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/41
Other Adverse Events (participants affected / at risk) | 2/8 | 1/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Case Group (N=8) | Control Group (N=41)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Shoulder joint repair (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes